CLINICAL TRIAL: NCT07250113
Title: WeCareToFeedDysphagia to Reduce Care-partner Burden Full-scale RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Liron Sinvani, Associate Professor, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 25-0388; R33AG079930 (NIH)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Caregiver Burden; Alzheimer's Disease; Dementia; Oropharyngeal Dysphagia; Older Adults
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease; Dementia; Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Control + WeCareToFeedDysphagia (Experimental): Participants receive usual care from their medical team and receive contact information for speech-language pathology follow-up care. Participants will also receive access to the WeCareToFeedDysphagia web tool and receive text message reminders to use the tool.
  Interventions: Behavioral: WeCareToFeedDysphagia web tool
- Enhanced Control (No Intervention): Participants receive usual care from their medical team and receive contact information for speech-language pathology follow-up care.

INTERVENTIONS:
Behavioral: WeCareToFeedDysphagia web tool — The web tool uses written and video content, care-partner testimonials, frequently asked questions, and resource links to provide accurate information (e.g., dysphagia diets), set realistic expectations, identify/support feeding goals (quality of life considerations), acknowledge/support care-partner feelings, and provide competencies/skills for oropharyngeal dysphagia (OD) management.
  Arms: Enhanced Control + WeCareToFeedDysphagia

SUMMARY:
The goal of this clinical trial is to learn if a newly-created website tool, called WeCareToFeedDysphagia, helps to reduce feelings of burden in care partners of patients with Alzheimer's disease and related dementias (AD/ADRD) who were diagnosed with trouble swallowing (oropharyngeal dysphagia). The main questions this study aims to answer are:

* How effective is the WeCareToFeedDysphagia tool in reducing feelings of burden in care partners?
* Does the WeCareToFeed Dysphagia tool help improve patient outcomes?
* Does care partner age, gender, and patient dysphagia severity impact the strength of the effect of the WeCareToFeedDysphagia tool?
* Is the strength of the effect of the WeCareToFeedDysphagia tool impacted by care partner's beliefs in being able to manage behavior and stress (self-efficacy)?

Researchers will compare a group of care partners who have access to the WeCareToFeedDysphagia tool (intervention) to a group of care partners who do not have access to the tool. Both groups will receive contact information for help from a speech language pathologist expert (enhanced usual care).

Participants will:

* be given access to the web tool and receive 3 text message reminders over 3 weeks to use the tool (intervention group only).
* be asked to complete a remote, web-based survey three times: when enrolled in the study, at 1 month following patient leaving the hospital, and at 3 months following patient leaving the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as the primary care partner of an older adult patient (patient age ≥ 65 years) with AD/ADRD and oropharyngeal dysphagia (OD) admitted to the Northwell medicine service
* Age ≥ 18 years
* Designated as the legally authorized representative (LAR) or health care proxy (HCP), or designated by the LAR or HCP to participate
* Proficient in English
* Has access to a device (e.g. smartphone, iPad, computer) capable of accessing a web browser

Exclusion Criteria:

* Care partner of patient with a percutaneous feeding tube (i.e. PEG, PEJ used exclusively)
* Care partner of patient who will not be discharged to the home or community setting (e.g., home, assisted living, independent living)
* Care partner will not be involved with OD management (e.g. buying or making food, feeding, supervising) after hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Mean Care Partner Burden at 3 Months Post Hospital Discharge | 3 months from hospital discharge
  Burden will be measured using the Zarit Burden Scale (ZBI-22), a validated measure that assesses 22 statements related to personal strain accompanying caring for another person, which is rated with 5 frequency-related response categories, scored 0 (never) to 4 (nearly always). The total score ranges between 0 and 88 (higher scores indicating higher burden). A score greater than 21 has been suggested to indicate care-partner burden. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.

SECONDARY OUTCOMES:
Mean Care Partner Burden at 1 Month Post Hospital Discharge | 1 month from hospital discharge
  Burden will be measured using the Zarit Burden Scale (ZBI-22), a validated measure that assesses 22 statements related to personal strain accompanying caring for another person, which is rated with 5 frequency-related response categories, scored 0 (never) to 4 (nearly always). The total score ranges between 0 and 88 (higher scores indicating higher burden). A score greater than 21 has been suggested to indicate care-partner burden. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean Care Partner Quality of Life at 1 Month Post Hospital Discharge | 1 month from hospital discharge
  Care Partner Quality of Life (CarerQol) will be measured using the validated Care-Related Qol-7D. The Care-Related Qol-7D measures well-being (CarerQol-VAS or visual analog scale) and subjective burden. The CarerQol-VAS measures happiness, using endpoints between 'completely unhappy' (0) and 'completely happy' (10). Subjective burden is measured on 7 dimensions (fulfillment, relational problems, mental health, daily activities problems, physical health, and support), and rated as (i) no, (ii) some, and (iii) a lot. The weighted score ranges from 0-100 (worst to best caregiving situation). Higher scores indicate higher quality of life. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean Care Partner Quality of Life at 3 Months Post Hospital Discharge | 3 months from hospital discharge
  Care Partner Quality of Life (CarerQol) will be measured using the validated Care-Related Qol-7D. The Care-Related Qol-7D measures well-being (CarerQol-VAS or visual analog scale) and subjective burden. The CarerQol-VAS measures happiness, using endpoints between 'completely unhappy' (0) and 'completely happy' (10). Subjective burden is measured on 7 dimensions (fulfillment, relational problems, mental health, daily activities problems, physical health, and support), and rated as (i) no, (ii) some, and (iii) a lot. The weighted score ranges from 0-100 (worst to best caregiving situation). Higher scores indicate higher quality of life. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Percent Engagement with the WeCareToFeedDysphagia Tool | 3 months from hospital discharge
  Engagement with WeCareToFeedDysphagia will be defined as percent of care partners viewing 2 or more pages within the tool. Success will be defined as greater than or equal to 45% of care partners engaging with the tool. Data will be captured via Google Analytics data to assess program usage in the domains of time/date of login, duration of page views, and document downloaded Engagement with the tool will be reported for the intervention arm only.

OTHER OUTCOMES:
Mean CARES Part A at 1 Month Post Hospital Discharge | 1 month from hospital discharge
  The Caregiver Analysis of Reported Experiences with Swallowing Disorders (CARES) Part A Checklist of Behavioral Changes is a 10-item questionnaire that measures responses to yes/no statements. Part A is scored 1 point for every yes response out of a maximum of 10 points. Scores are continuous, with lower scores indicating more self-efficacy with behavioral management. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean CARES Part A at 3 Months Post Hospital Discharge | 3 months from hospital discharge
  The Caregiver Analysis of Reported Experiences with Swallowing Disorders (CARES) Part A Checklist of Behavioral Changes is a 10-item questionnaire that measures responses to yes/no statements. Part A is scored 1 point for every yes response out of a maximum of 10 points. Scores are continuous, with lower scores indicating more self-efficacy with behavioral management. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean CARES Part B at 1 Month Post Discharge | 1 month from hospital discharge
  The Caregiver Analysis of Reported Experiences with Swallowing Disorders (CARES) Part B Measures of Subjective Caregiver Stress is a 16-item questionnaire that measures responses to yes/no statements. Part B is scored 1 point for every yes response out of a maximum of 16 points. Scores are continuous, with lower scores indicating more self-efficacy with stress management. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean CARES Part B at 3 Months Post Hospital Discharge | 3 months from hospital discharge
  The Caregiver Analysis of Reported Experiences with Swallowing Disorders (CARES) Part B Measures of Subjective Caregiver Stress is a 16-item questionnaire that measures responses to yes/no statements. Part B is scored 1 point for every yes response out of a maximum of 16 points. Scores are continuous, with lower scores indicating more self-efficacy with stress management. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean EdFED-Q at 1 Month Post Hospital Discharge | 1 month from hospital discharge
  The Edinburgh Feeding Evaluation in Dementia Questionnaire (EdFED-Q) is an 11-item instrument which assesses eating and feeding problems in people with late-stage dementia. The care partner assigns a score (0 to 2, never, sometimes, or often occurring) to each item; higher scores (maximum of 20) indicate greater feeding dysfunction. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean EdFED-Q at 3 Months Post Hospital Discharge | 3 months from hospital discharge
  The Edinburgh Feeding Evaluation in Dementia Questionnaire (EdFED-Q) is an 11-item instrument which assesses eating and feeding problems in people with late-stage dementia. The care partner assigns a score (0 to 2, never, sometimes, or often occurring) to each item; higher scores (maximum of 20) indicate greater feeding dysfunction. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean QUALID at 1 Month Post Hospital Discharge | 1 month from hospital discharge
  The Quality of Life in Late-Stage Dementia Scale (QUALID) is an 11 item, validated scale administered to care partners for rating quality of life in late stage dementia. A 5 point scale (1-5) is used to capture the frequency of each item. Scores range from 11 to 55, with lower scores reflecting a higher quality of life. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean QUALID at 3 Months Post Hospital Discharge | 3 months from hospital discharge
  The Quality of Life in Late-Stage Dementia Scale (QUALID) is an 11 item, validated scale administered to care partners for rating quality of life in late stage dementia. A 5 point scale (1-5) is used to capture the frequency of each item. Scores range from 11 to 55, with lower scores reflecting a higher quality of life. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean Patient Acute Care Visits at 1 Month Post Hospital Discharge | 1 month from hospital discharge
  Care partners will be asked to report acute care visits defined as emergency department visits and hospital readmissions for the patient they care for. Visits will be distinguished as aspiration-related or non-aspiration related complaints and reported as yes (took place) or no (did not take place). More frequently reported acute care visits will be associated with worse patient outcomes. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean Patient Acute Care Visits at 3 Months Post Hospital Discharge | 3 months from hospital discharge
  Care partners will be asked to report acute care visits defined as emergency department visits and hospital readmissions for the patient they care for. Visits will be distinguished as aspiration-related or non-aspiration related complaints and reported as yes (took place) or no (did not take place). More frequently reported acute care visits will be associated with worse patient outcomes. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean Patient Dehydration Events at 1 Month Post Hospital Discharge | 1 month from hospital discharge
  Care partners will be asked to report dehydration events requiring intravenous or subcutaneous fluid administration for the patient they care for as yes (took place) or no (did not take place). More dehydration events will be associated with worse outcomes. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean Patient Dehydration Events 3 Months Post Hospital Discharge | 3 months from hospital discharge
  Care partners will be asked to report dehydration events requiring intravenous or subcutaneous fluid administration for the patient they care for as yes (took place) or no (did not take place). More dehydration events will be associated with worse outcomes. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean Patient Weight Loss 1 Month Post Hospital Discharge | 1 month from hospital discharge
  Caregivers will be asked to report patient weight loss via a single-item question derived from the Mini Nutritional Assessment (MNA). Results will be averaged and categorized as weight loss greater than 3 kg, weight loss 1-3 kg, and no weight loss. More weight loss will be associated with worse outcomes. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean Patient Weight Loss 3 Months Post Hospital Discharge | 3 months from hospital discharge
  Caregivers will be asked to report patient weight loss via a single-item question derived from the Mini Nutritional Assessment (MNA). Results will be averaged and categorized as weight loss greater than 3 kg, weight loss 1-3 kg, and no weight loss. More weight loss will be associated with worse outcomes. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean NPI-Q 1 Month Post Hospital Discharge | 1 month from hospital discharge
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) is a validated tool with 12 behavioral domains for the assessment of neuropsychiatric symptomology designed for completion by caregivers of patients with Alzheimer's Disease and Related Dementias. The tool asks the interviewee to rate each symptom, if present, as mild, moderate, or severe. Total scores range from 0-36 with higher scores indicating greater prominence of dementia symptoms. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.
Mean NPI-Q 3 Months Post Hospital Discharge | 3 months from hospital discharge
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) is a validated tool with 12 behavioral domains for the assessment of neuropsychiatric symptomology designed for completion by caregivers of patients with Alzheimer's Disease and Related Dementias. The tool asks the interviewee to rate each symptom, if present, as mild, moderate, or severe. Total scores range from 0-36 with higher scores indicating greater prominence of dementia symptoms. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message.

CONTACTS AND LOCATIONS:
Overall Officials: Liron Sinvani, MD, Principal Investigator — Northwell Health

IPD SHARING:
Plan to Share IPD: Yes
All data which can be sufficiently deidentified to preserve participant confidentiality will be made available via the Open Science Framework (OSF) repository. The goal of all shared data will be to facilitate replication of all primary and secondary, and exploratory study analyses as well as to allow for additional analyses with available data. Data will be redacted according to the safe-harbor method, and effective strategies will be adopted to minimize risk of disclosing a participant's identity. Data will be shared along with documentation of how variables were cleaned, coded, or summarized. In cases where participant-level data could be used to identify individuals, summary data will be presented (e.g. presenting an age category ">85 years old" rather than individual participant age). Information about how summary data was generated will be provided in the data dictionary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data and metadata will be available in advance of the first online publication of the primary study outcomes. De-identified data will be stored on OSF indefinitely to allow for continued access.
Access Criteria: Deidentified data will be made publicly available.